CLINICAL TRIAL: NCT07010640
Title: A Comparison of Video Versus Written Instructions for Early Motion Flexors Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 240624458
Record Dates: First submitted 2025-02-19; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Compliance, Treatment; Hand Flexor Repair; Compliance to Rehabilitation After Hand Flexor Repair
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: One group of participants will receive written instructions following hand flexor repair, whilst the other group will receive video instructions in addition to written on instructions.
Who Masked: Participant
Masking Description: Participants will be informed that they are taking part in a study, but no distinction will be made between written and video instructions. Participants receiving written instructions will not be made aware of the alternative video instructions. Similarly, participants receiving video instructions will not be made aware that they are part of the experimental group and that the other group is not receiving video instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Instructions Group (Experimental): In addition to written instructions, will receive video instructions to facilitate rehabilitation process.
  Interventions: Other: Video Instrctions
- Written Instructions Group (No Intervention): Will only receive written instructions for rehabilitation process.

INTERVENTIONS:
Other: Video Instrctions — Video instructions of rehabilitation techniques and movements to help with adherence and compliance to treatment.
  Arms: Video Instructions Group

SUMMARY:
The research objective is to evaluate the efficacy of video instructions compared to written or verbal instructions for early motion rehabilitation following hand flexor repair. The primary research question addresses whether video instructions improve compliance with early motion rehabilitation post-surgery compared to traditional methods. The hypothesis is that patients who receive video instructions are more likely to adhere to their rehabilitation regimen than those who receive verbal or written instructions.

DETAILED DESCRIPTION:
Flexor tendon injuries are prevalent, particularly among the working-age population, leading to significant disability and financial burden, with annual costs ranging from $240 to $409 million in the United States. Effective rehabilitation is crucial to prevent complications like stiffness and adhesions. Advances in surgical techniques, such as multi-strand core sutures, have enabled early active rehabilitation. Previous studies indicate the benefits of video-assisted therapy and education in various medical contexts, suggesting that video instructions could similarly enhance compliance and outcomes in hand flexor rehabilitation. The study aims to assess the efficacy of video instructions versus written or verbal instructions for early motion rehabilitation following hand flexor repair.

The study consists of a single-center single-blinded randomized control trial comparing the communication methods of instructions for early motion rehabilitation following hand flexor repairs. All procedures will be performed under Wide-Awake Local Anesthesia No Tourniquet (WALANT). The sample size will consist of 60 participants. The subjects will be randomly assigned (1:1 randomization) to one of two groups; the experimental group will receive video instructions, while the control group written and verbal instructions. Both groups will be surgically managed by two board-certified orthopaedic hand surgeons (i.e., Christian Foy, MD & Eric Astacio, MD) at a supra-tertiary local hospital (i.e., Oncologic Hospital) under the same operative approach (i.e., six-strand flexor repair). All the subjects will receive the standard of care including a dorsal blocking splint and follow-up visits in hand clinic.

Data collection methods include: surveys, questionnaires (i.e., three - patient satisfaction, pain levels, and self-efficacy), clinical assessments (i.e., ROM, grip strength and complication rates), and communication with the therapist to assess exercise adherence and frequency.

The statistical analysis plan for this study involves summarizing the baseline characteristics of the study population and primary/secondary outcomes using descriptive statistics. Chi-square will be used to compare bivariate categorical variables while t-test will be used to analyze continuous non-parametric variables. A multivariate analysis will be used to control for potential confounder and assess the independent effect of the instruction method on outcomes. A 95% confidence interval with an alpha of 0.05 will be considered statistically significant. Microsoft Excel and STATA software will be used for statistical analysis.

A waiver from the IRB will be requested to gain authorization for the release of health information. All patient records will be kept under use for the duration of the study. The estimated duration of this study is 1 year.

To protect patient confidentiality, data will be stored in an encrypted database in the orthopedic surgery department at the University of Puerto Rico (UPR) Medical Sciences Campus. Only study personnel will have access to the room and computer where digital files will be stored. The information will be coded with identification numbers, and the data will be stored using only these numbers. The information that will be obtained from this study will be used for the purpose specified in the protocol, and the identity of the patients will not be traced after coding. The study will be approved by the proposed research performance site Institutional Review Board (IRB) prior to the initiation of the study. No subjects will be identified by name, social security number, or any other HIPAA identifier in any reports. Any incident regarding information security and/or privacy will be reported in accordance with University Hospital/Medical Sciences Campus policy and procedures in place for reporting incidents, i.e. theft or loss of data or storage media, unauthorized access of sensitive data or storage devices or non-compliance with security controls.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years old or older Isolated flexor injuries Procedures performed under WALANT technique Providing written informed consent

Exclusion Criteria:

Patients younger than 18 years old Patients with other injuries Procedures performed under any anesthesia other than WALANT Mental disability History of psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Range of motion (i.e., using a goniometer)
Patient-reported outcomes | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Visual Analog Scale (VAS) Measuring distance from 1-100 millimeters. Higher scores indicate pain, whilst lower scores indicate less or no pain.
Compliance with Rehabilitation Protocol | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Frequency of the early motion exercises (i.e., track how often the patients perform their rehabilitation exercises)
Functional Outcome | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Grip strength (i.e., using a dynamometer)
Patient Reported Outcomes | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Numeric Rating Scale (NRS) A ten point scale, with 0 representing no pain and 10 representing the worst possible pain.
Patient Reported Outcomes | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Disabilities of the Arm, Shoulders and Hand (DASH) A self report questionnaire, scored from 0-100. Higher scores indicate a more severe disability, lower scores indicate little or no disability.
Patient Reported Outcomes | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Patient Rated Wrist Evaluation (PRWE) Patient rate their pain and disabilities using wrist over the last week, on a score from 0-10. Higher scores indicate a higher degree of pain and disability.
Patient Reported Outcomes | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Satisfaction with instruction methods: utilize a standardized questionnaire to gauge patient satisfaction with the instruction method (i.e., the system usability scale or a custom satisfaction survey)
Compliance with Rehabilitation Protocol | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Adherence to physical therapy (i.e., via self-reports or therapist assessments)
Compliance with Rehabilitation Protocol | The measurement is assessed at 2 weeks, 6 weeks, and 3 months.
  Duration of the early motion exercises (i.e., track for how long the patients perform their rehabilitation exercises)

SECONDARY OUTCOMES:
Clinical outcomes | 3 months after surgery
  Complication rates: track the incidence of adhesions, re-ruptures, and infections.
Rehabilitation efficiency | 3 months after surgery
  Number of follow-up visits: compare the number of follow-up visits required for each group.
Cognitive outcome | 3 months after surgery
  Instruction comprehension: assess the understanding of the instructions through a quiz or verbal feedback.
Clinical Outcomes | 3 months after surgery
  Time to return to work: measure the time taken for patients to return to their usual activities or work.
Cognitive Outcome | 3 months after surgery
  Self-efficacy: use the general Self-Efficacy Scale to measure the patient's confidence in performing their rehabilitation exercises.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Foy, M.D., Principal Investigator — Orthopaedic Surgery Department, School of Medicine
Locations (2):
- Puerto Rico (2):
  - Orthopaedic Surgery Clinic at ASEM, San Juan, PR
  - Puerto Rico Level 1 Trauma Hospital, San Juan, PR

IPD SHARING:
Plan to Share IPD: No